CLINICAL TRIAL: NCT02314702
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® L Revision Femoral Stems
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002L
Record Dates: First submitted 2014-12-03; First posted 2014-12-11 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Joint Disease
Keywords: Osteoarthritis; Avascular necrosis; Ankylosis; Protrusio acetabuli; Painful hip dysplasia; Rheumatoid arthritis; Correction of functional deformity; Revision procedures
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Revision Total Hip Arthroplasty: Single study group previously implanted with a PROFEMUR® L Revision Femoral Stem
  Interventions: Device: PROFEMUR® L Revision Femoral Stem

INTERVENTIONS:
Device: PROFEMUR® L Revision Femoral Stem — Revision Total Hip Arthroplasty
  Other Names: Hip Revision Device

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this PMCF study to evaluate the safety and efficacy of its THA and resurfacing components marketed in the EU. These types of studies are required by regulatory authorities for all THA and resurfacing devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with MEDDEV 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone revision total hip arthroplasty
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Exclusion Criteria:

* Subjects currently enrolled in another clinical study
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or have pending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with PROFEMUR® L Revision Femoral Components
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants who require a revision | 10 years post-operative
  The primary objective of this study is to estimate the revision rate of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional score on the the Oxford Hip Score instrument | Screening (First Available), 2-5 years, 5-7 years, and 10 years
  To characterize patient hip-related health status, as assessed by Oxford Hip Scores
Patient functional score on the EQ-5D-3L instrument | Screening (First Available), 2-5 years, 5-7 years, and 10 years
  To characterize patient general health status, as assessed by EQ-5D-3L scores

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No